CLINICAL TRIAL: NCT04732117
Title: A Randomized, Double-blind, Placebo Controlled, Multicenter, Phase III Study of Subcutaneous Secukinumab to Compare Efficacy at 16 Weeks With Placebo and to Assess Safety and Tolerability up to 52 Weeks in Chinese Participants With Active Non-radiographic Axial Spondyloarthritis
Brief Title: Efficacy and Safety Study of Secukinumab in Chinese Participants With Non-radiographic Axial Spondyloarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457I2301
Record Dates: First submitted 2021-01-28; First posted 2021-02-01 (Actual); Results first posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Non-radiographic Axial Spondyloarthritis
Keywords: non-radiographic spondyloarthritis; chronic inflammatory disease; inflammatory back pain,; secukinumab; AIN457
MeSH Terms: conditions — Non-Radiographic Axial Spondyloarthritis | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Secukinumab (Experimental): Participants received secukinumab 150 mg in a pre-filled syringe (PFS). Treatment was double-blinded until Week 12. From Week 16, participants continued with an open-label treatment of secukinumab 150 mg. At Week 24, non-responders (not achieving ASAS20) were escalated to secukinumab 300 mg, while responders continued with secukinumab 150 mg.
  Interventions: Drug: Secukinumab
- Placebo (Placebo Comparator): Participants initially received a placebo in a pre-filled syringe (PFS) in a double-blinded manner until Week 12. At Week 16, they switched to an open-label treatment of secukinumab 150 mg. At Week 24, non-responders (not achieving ASAS20) were escalated to secukinumab 300 mg, while responders continued with secukinumab 150 mg.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Secukinumab — Secukinumab 150 mg s.c. using a PFS at Baseline, Weeks 1, 2, and 3, followed by administration every 4 weeks from Week 4 until Week 12. At Week 16, all participants continued or switched to receiving secukinumab 150 mg s.c. every 4 weeks, using a PFS. This treatment regimen continued from Week 16 through Week 48. For participants who did not respond to the secukinumab 150 mg dose during the open-label period, the dose was increased to 300 mg s.c., using two PFS, also administered every 4 weeks.
  Other Names: AIN457
  Arms: Secukinumab
Drug: Placebo — Placebo s.c. using a PFS at baseline, Weeks 1, 2 and 3, followed by administration every 4 weeks from Week 4 until Week 12.
  Arms: Placebo

SUMMARY:
The purpose of this study was to evaluate the efficacy, safety, and tolerability of secukinumab in Chinese patients with active non-radiographic axial spondyloarthritis (nr-axSpA).

DETAILED DESCRIPTION:
This was a randomized, double-blind, placebo-controlled study. Approximately 134 participants were planned to be randomized in a 1:1 ratio to receive secukinumab 150 mg subcutaneously (s.c.) or placebo.

The double-blind treatment period lasted for 16 weeks. At the end of this period, all participants, including those who initially received placebo, switched to open-label treatment with secukinumab 150 mg s.c.

The first dose of open-label treatment was administered at the Week 16 visit, after completing all necessary assessments for that visit. However, the participants and investigators remained blinded to the original treatment assignment. At Week 24, participants who did not respond to the treatment (defined as not achieving Ankylosing SpondyloArthritis International Society 20 [ASAS20] response) were given a higher dose of secukinumab (300 mg s.c.), while responders continued with the 150 mg s.c. dose. The study treatment continued until Week 48. Four weeks after the last study treatment administration, an end-of-treatment visit was conducted at Week 52.

Additionally, a post-treatment safety follow-up visit was performed 12 weeks after the last study treatment administration for all participants, whether they completed the entire study as planned or exited early.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-nursing female patients at least 18 years of age
* Diagnosis of axial spondyloarthritis according to Ankylosing SpondyloArthritis International Society (ASAS) axial spondyloarthritis criteria
* Objective signs of inflammation (magnetic resonance imaging (MRI) or abnormal C-reactive protein)
* Active axial spondyloarthritis as assessed by total Bath Ankylosing Spondylitis Disease Activity Index >=4 cm
* Spinal pain as measured by Bath Ankylosing Spondylitis Disease Activity Index question #2 ≥ 4 cm (0-10 cm) at baseline
* Total back pain as measured by Visual Analogue scale ≥ 40 mm (0-100 mm) at baseline
* Patients should have been on at least 2 different non-steroidal anti-inflammatory drugs with an inadequate response
* Patients who have been on a TNFα inhibitor (not more than one) must have experienced an inadequate response

Exclusion Criteria:

* Patients with radiographic evidence for sacroiliitis, grade ≥ 2 bilaterally or grade ≥ 3 unilaterally
* Inability or unwillingness to undergo MRI
* Chest X-ray or MRI with evidence of ongoing infectious or malignant process
* Patients taking high potency opioid analgesics
* Previous exposure to secukinumab or any other biologic drug directly targeting interleukin-17 (IL-17) or IL-17 receptor
* Pregnant or nursing (lactating) women

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2025-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (24):
- China (24):
  - Novartis Investigative Site, Hefei, Anhui
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Xiamen, Fujian
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Shantou, Guangdong
  - Novartis Investigative Site, Shenzhen, Guangdong
  - Novartis Investigative Site, Harbin, Heilongjiang
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Baotou, Inner Mongolia
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Yangzhou, Jiangsu
  - Novartis Investigative Site, Nanchang, Jiangxi
  - Novartis Investigative Site, Pingxiang, Jiangxi
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Linyi, Shandong
  - Novartis Investigative Site, Ürümqi, Xinjiang
  - Novartis Investigative Site, Kunming, Yunnan
  - Novartis Investigative Site, Ningbo, Zhejiang
  - Novartis Investigative Site, Wenzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Bengbu
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A screening period of up to 10 weeks before randomization assessed participant eligibility
Groups:
- Placebo: Participants initially received placebo in a pre-filled syringe (PFS) in a double-blinded manner until Week 12. At Week 16, they switched to an open-label treatment of secukinumab 150 mg. At Week 24, non-responders (not achieving ASAS20) were escalated to secukinumab 300 mg, while responders continued with secukinumab 150 mg.
Period: Double-Blind period (up to Week 16)
Arm/Group | Secukinumab | Placebo
Started | 68 | 69
Completed | 67 | 68
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Subject Decision | 0 | 1
Period: Open-label period
Arm/Group | Secukinumab | Placebo
Started | 67 | 68
Escalated to secukinumab 300 mg (Participants who were non-responders at Week 24 and escalated to secukinumab 300 mg) | 12 | 17
Completed | 64 | 65
Not Completed | 3 | 3
Not completed — Subject discontinuation | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Secukinumab | Placebo | Total
Number analyzed (Participants) | 68 | 69 | 137
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.4 (7.83) | 29.4 (7.44) | 29.4 (7.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 17 | 40
  Male | 45 | 52 | 97
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 68 | 69 | 137
TNF-alpha inhibitors exposure [Count of Participants; unit: Participants]
  TNF alpha-inhibitor-naive | 61 | 62 | 123
  Prior exposure to a TNF-alpha inhibitor | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Assessment of SpondyloArthritis International Society 40 (ASAS40) Response Rate in TNF-alpha-inhibitor-naive Participants at Week 16
Description: ASAS40 response was defined as relative improvement of at least 40% and absolute improvement of at least 2 units on a 0 to 10 scale in at least 3 of the 4 main domains of the ASAS and no worsening at all in the remaining domain.
  The 4 main domains of the ASAS are: 1.Patient's Global Assessment of Disease Activity (score ranged from 0 [not active] to 10 [very active]); 2.Back Pain (score ranged from 0 [no pain] to 10 [severe pain]); 3.Function (Bath Ankylosing Spondylitis Functional Index [BASFI]) (score ranged from 0 [easy] to 10 [impossible]); 4.Inflammation (mean of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) questions 5 and 6 concerning morning stiffness intensity and duration) (score ranged from 0 [none] to 10 [very severe]).
  The percentage of TNF-alpha-inhibitor-naïve participants who achieved ASAS40 response at Week 16 was assessed using a logistic regression model. Discontinued participants and those with missing responses were considered non-responders
Time Frame: Baseline, Week 16
Population: All randomized participants to whom study treatment was assigned and who were TNF-alpha-naive at baseline
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 61 | 62
Percentage of participants | 58.72 [46.41 to 71.03] | 26.03 [15.12 to 36.94]

2. Secondary Outcome: ASAS40 Response Rate in All Participants at Week 16
Description: ASAS40 response was defined as relative improvement of at least 40% and absolute improvement of at least 2 units on a 0 to 10 scale in at least 3 of the 4 main domains of the ASAS and no worsening at all in the remaining domain.
  The 4 main domains of the ASAS are: 1.Patient's Global Assessment of Disease Activity (score ranged from 0 [not active] to 10 [very active]); 2.Back Pain (score ranged from 0 [no pain] to 10 [severe pain]); 3.Function (BASFI) (score ranged from 0 [easy] to 10 [impossible]); 4.Inflammation (mean of BASDAI questions 5 and 6 concerning morning stiffness intensity and duration) (score ranged from 0 [none] to 10 [very severe]).
  The percentage of participants who achieved ASAS40 response at Week 16 was assessed using a logistic regression model. Discontinued participants and those with missing responses were considered non-responders
Time Frame: Baseline, Week 16
Population: All randomized participants to whom study treatment was assigned
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 68 | 69
Percentage of participants | 60.10 [48.46 to 71.75] | 24.78 [14.57 to 34.98]

3. Secondary Outcome: ASAS 5/6 Response Rate at Week 16.
Description: The ASAS 5/6 response was defined as an improvement of ≥20% in at least five of all six domains of the ASAS: 1.Patient's Global Assessment of Disease Activity (score ranged from 0 [not active] to 10 [very active]); 2.Back Pain (score ranged from 0 [no pain] to 10 [severe pain]); 3.Function (BASFI) (score ranged from 0 [easy] to 10 [impossible]); 4.Inflammation (mean of BASDAI questions 5 and 6 concerning morning stiffness intensity and duration) (score ranged from 0 [none] to 10 [very severe]); 5) spinal mobility represented by the BAS Disease Metrology Index (BASDMI) (scale ranged from 0 [no limitation of movement] to 10 [very severe limitation of movement]; and 6) C-reactive protein (acute phase reactant).
  The percentage of participants who achieved ASAS 5/6 response at Week 16 was assessed using a logistic regression model. Missing responses were imputed as non-responders. Discontinued participants were considered non-responders
Time Frame: Baseline, Week 16
Population: All randomized participants to whom study treatment was assigned
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 68 | 69
Percentage of participants | 61.97 [51.12 to 72.82] | 25.89 [16.13 to 35.64]

4. Secondary Outcome: Change From Baseline in Total Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Score at Week 16
Description: The BASDAI consisted of a 0 through 10 scale (0 being no problem and 10 being the worst problem, captured as a continuous VAS), which was used to answer 6 questions pertaining to the 5 major symptoms of AS: 1. Fatigue; 2. Spinal pain; 3. Joint pain / swelling; 4. Areas of localized tenderness (called enthesitis, or inflammation of tendons and ligaments); 5. Morning stiffness duration; 6. Morning stiffness severity. BASDAI score was calculated as the mean of the questions 5 and 6. The resulting 0 to 10 score was added to the scores from questions 1-4. The resulting 0 to 50 score was divided by 5 to give a final 0-10 BASDAI score, where higher score indicated high disease activity.
  The change from baseline in BASDAI scores at Week 16 was assessed using Mixed-effects model repeated measures (MMRM). A negative change from baseline indicated improvement.
Time Frame: Baseline, Week 16
Population: All randomized participants to whom study treatment was assigned with measures at both baseline and Week 16
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 66 | 65
Score on a scale | -3.70 (0.240) | -2.15 (0.237)

5. Secondary Outcome: BASDAI 50 Rate at Week 16
Description: The BASDAI consisted of a 0 through 10 scale (0 being no problem and 10 being the worst problem, captured as a continuous VAS), which was used to answer 6 questions pertaining to the 5 major symptoms of AS: 1. Fatigue; 2. Spinal pain; 3. Joint pain / swelling; 4. Areas of localized tenderness (called enthesitis, or inflammation of tendons and ligaments); 5. Morning stiffness duration; 6. Morning stiffness severity. BASDAI score was calculated as the mean of the questions 5 and 6. The resulting 0 to 10 score was added to the scores from questions 1-4. The resulting 0 to 50 score was divided by 5 to give a final 0-10 BASDAI score, where higher score indicated high disease activity. BASDAI 50 was defined as an improvement of at least 50% in the BASDAI total score compared to baseline.
  The percentage of participants achieving BASDAI 50 at Week 16 was assessed using a logistic regression model. Discontinued participants and with missing responses were considered non-responders
Time Frame: Baseline, Week 16
Population: All randomized participants to whom study treatment was assigned
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 68 | 69
Percentage of participants | 64.04 [52.82 to 75.27] | 25.77 [15.68 to 35.85]

6. Secondary Outcome: Change From Baseline of High Sensitivity C-Reactive Protein (hsCRP) at Week 16
Description: hsCRP was measured as a marker of inflammation from blood samples. The change from baseline in hsCRP at Week 16 was assessed using MMRM. It was expressed as a ratio of Week 16 to baseline values. Ratios less than 1.0 at Week 16 represented reduced hsCRP.
Time Frame: Baseline, Week 16
Population: All randomized participants to whom study treatment was assigned with measures at both baseline and Week 16
Measure: Least Squares Mean (Standard Error); unit: Ratio: Week 16 / Baseline
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 64 | 65
Ratio: Week 16 / Baseline | 0.38 (1.137) | 0.74 (1.136)

7. Secondary Outcome: Change From Baseline in Total Bath Ankylosing Spondylitis Functional Index (BASFI) at Week 16
Description: The BASFI is a set of 10 questions designed to determine the degree of functional limitation in subjects with AS. The questions were chosen on the basis of predominant input from subjects with AS. The first eight questions consider activities related to functional anatomy. The final two questions assess the subjects' ability to cope with everyday life. A 0-10 scale (captured as a continuous VAS) is used to answer the questions. The BASFI score is the mean of the ten scales - a value between 0 and 10, with higher scores indicating a higher degree of functional limitation in patients. The change from baseline in BASFI at Week 16 was assessed. A negative change from baseline indicated improvement.
Time Frame: Baseline, Week 16
Population: All randomized participants to whom study treatment was assigned with measures at both baseline and Week 16
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 66 | 65
Score on a Scale | -2.04 (0.225) | -0.93 (0.222)

8. Secondary Outcome: Change From Baseline in Sacroiliac Joint (SIJ) Edema Score on Magentic Resonance Imaging (MRI) at Week 16
Description: The MRI assessment of the total edema score of the Sacroiliac Joint (SIJ) measured the degree of edema or fluid accumulation in the joint. The score ranged from 0 to 24, with higher scores indicating more severe inflammation. The change from baseline in inflammation, as measured by the SI joint total edema score at Week 16, was evaluated using an ANCOVA model. Any missing data was imputed using multiple imputation prior to running the ANCOVA analysis.
Time Frame: Baseline, Week 16
Population: All randomized participants to whom study treatment was assigned with measures at both baseline and Week 16
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 65 | 66
Score on a Scale | -3.09 (0.34) | -0.84 (0.35)

9. Secondary Outcome: ASAS20 Response Rate at Week 16
Description: ASAS20 response was defined as relative improvement of at least 20% and absolute improvement of at least 1 unit on a 0 to 10 scale in at least 3 of the 4 main domains of the ASAS and no worsening of ≥20% and ≥1 unit at all in the remaining domain.
  The 4 main domains of ASAS are 1.Patient's Global Assessment of Disease Activity (score ranged from 0 [not active] to 10 [very active]); 2.Back Pain (score ranged from 0 [no pain] to 10 [severe pain]); 3.Function (BASFI) (score ranged from 0 [easy] to 10 [impossible]); 4.Inflammation (mean of BASDAI questions 5 and 6 concerning morning stiffness intensity and duration) (score ranged from 0 [none] to 10 [very severe]) The percentage of participants who achieved ASAS20 response at Week 16 was assessed using a logistic regression model. Discontinued participants and those with missing responses were considered non-responders
Time Frame: Baseline, Week 16
Population: All randomized participants to whom study treatment was assigned
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 68 | 69
Percentage of participants | 78.10 [68.29 to 87.91] | 47.60 [35.82 to 59.39]

10. Secondary Outcome: Change From Baseline in Short Form-36 Physical Component Summary (SF-36 PCS) at Week 16
Description: SF-36 was an instrument used to measure health-related quality of life among healthy patients and patients with acute and chronic conditions. It consisted of eight subscales (domains) that could be scored individually: Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role- Emotional, and Mental Health. Each domain score ranged from 0 to 100, with higher scores indicating a higher level of functioning. The Physical Component Summary (PCS) was an overall summary score calculated from the 8 domains. It was a norm-based score with a mean of 50 and a standard deviation of 10. Higher scores indicated a higher level of functioning.
  The change from baseline in PCS at Week 16 was evaluated using MMRM. A positive change from baseline indicated an improvement.
Time Frame: Baseline, Week 16
Population: All randomized participants to whom study treatment was assigned with measures at both baseline and Week 16
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 67 | 67
Score on a Scale | 9.35 (0.772) | 4.34 (0.753)

11. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Quality of Life (ASQoL) Scores at Week 16
Description: The ASQoL was a self-administered questionnaire designed to assess health-related quality of life (HRQoL) in participants with ankylosing spondylitis. The ASQoL contained 18 items with a dichotomous yes/no response option. A single point was assigned for each "yes" response and no points for each "no" response resulting in overall scores that ranged from 0 (least severity) to 18 (highest severity). As such, a lower score indicated a better quality of life. Items included an assessment of mobility/energy, self-care, and mood/emotion.
  The change from baseline in ASQoL at Week 16 was assessed using MMRM. A negative change from baseline indicated an improvement.
Time Frame: Baseline, Week 16
Population: All randomized participants to whom study treatment was assigned with measures at both baseline and Week 16
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 67 | 67
Score on a scale | -4.90 (0.455) | -3.07 (0.447)

12. Secondary Outcome: ASAS Partial Remission Rate at Week 16
Description: The ASAS partial remission criteria were defined as a value not above 2 units (on a scale of 10) in each of the 4 main ASAS domains: 1. Patient's Global Assessment of Disease Activity (score ranged from 0 [not active] to 10 [very active]); 2. Back Pain (assessed on a scale of 0 [no pain] to 10 [severe pain]); 3. Function (BASFI) (score ranged from 0 [easy] to 10 [impossible]); 4. Inflammation (mean of BASDAI questions 5 and 6 concerning morning stiffness intensity and duration) (score ranged from 0 [none] to 10 [very severe]).
  The percentage of participants who achieved ASAS partial remission response at Week 16 was assessed using a logistic regression model. Missing responses were imputed as non-responders. Discontinued participants were considered non-responders.
Time Frame: Baseline, Week 16
Population: All randomized participants to whom study treatment was assigned
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 68 | 69
Percentage of participants | 30.83 [19.92 to 41.73] | 14.52 [6.23 to 22.80]

ADVERSE EVENTS:
Time Frame: From start of treatment to end of study, assessed up to approximately 65 weeks
Description: Any sign or symptom that occurred during the conduct of the trial
Groups:
- Secukinumab 150 mg: Participants who received at least one dose of secukinumab 150 mg during the 16-week double-blind treatment period or who received at least one dose of secukinumab 150 mg during the open- label treatment period. AEs were collected from the first dose of secukinumab 150 mg up to end of study or day of start of secukinumab 300 mg if dose escalation
- Secukinumab 300 mg: Participants who received at least one dose of secukinumab 300 mg during the open- label treatment period. AEs were collected from the first dose of secukinumab 300 mg up to end of study
- Any Secukinumab: Participants who received at least one dose of secukinumab, regardless of dose. AEs were collected from first dose of secukinumab up to end of study
- Placebo: Participants who received placebo. AEs were collected from first dose of placebo up to Week 16
Arm/Group | Secukinumab 150 mg | Secukinumab 300 mg | Any Secukinumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/135 | 0/29 | 0/135 | 0/69
Serious Adverse Events (participants affected / at risk) | 4/135 | 2/29 | 6/135 | 1/69
Other Adverse Events (participants affected / at risk) | 103/135 | 22/29 | 114/135 | 52/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab 150 mg (N=135) | Secukinumab 300 mg (N=29) | Any Secukinumab (N=135) | Placebo (N=69)
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Paronychia (Infections and infestations) | 0 | 1 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Neuroendocrine tumour of the rectum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Plasma cell mastitis (Reproductive system and breast disorders) | 1 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab 150 mg (N=135) | Secukinumab 300 mg (N=29) | Any Secukinumab (N=135) | Placebo (N=69)
Leukopenia (Blood and lymphatic system disorders) | 6 | 2 | 7 | 0
Monocytopenia (Blood and lymphatic system disorders) | 10 | 2 | 11 | 3
Diarrhoea (Gastrointestinal disorders) | 6 | 1 | 7 | 4
Pyrexia (General disorders and administration site conditions) | 7 | 1 | 8 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 6 | 1 | 7 | 2
Bronchitis (Infections and infestations) | 1 | 2 | 3 | 2
COVID-19 (Infections and infestations) | 23 | 4 | 27 | 7
Pharyngitis (Infections and infestations) | 3 | 3 | 5 | 1
Suspected COVID-19 (Infections and infestations) | 11 | 1 | 12 | 2
Tonsillitis (Infections and infestations) | 2 | 2 | 3 | 2
Upper respiratory tract infection (Infections and infestations) | 43 | 7 | 49 | 22
Urinary tract infection (Infections and infestations) | 9 | 1 | 10 | 4
Alanine aminotransferase increased (Investigations) | 11 | 1 | 12 | 5
Lipoprotein (a) increased (Investigations) | 4 | 0 | 4 | 5
Low density lipoprotein increased (Investigations) | 14 | 1 | 14 | 5
Weight increased (Investigations) | 4 | 2 | 6 | 0
White blood cells urine positive (Investigations) | 6 | 1 | 7 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 11 | 0 | 11 | 3
Hyperlipidaemia (Metabolism and nutrition disorders) | 23 | 0 | 23 | 10
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 9 | 1 | 10 | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 26 | 4 | 28 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 4 | 9 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 4 | 10
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 14 | 1 | 15 | 0
Proteinuria (Renal and urinary disorders) | 3 | 2 | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2020-11-16): https://cdn.clinicaltrials.gov/large-docs/17/NCT04732117/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-08): https://cdn.clinicaltrials.gov/large-docs/17/NCT04732117/SAP_001.pdf